CLINICAL TRIAL: NCT02229773
Title: Pharmacodynamics, Preliminary Pharmacokinetics and Tolerability After Multiple Oral Doses of 0.25 mg, 0.5 mg and 1 mg o.d. BIBB 1464 (Tablet) or Pravastatin 20 mg Over 2 Weeks in Hyperlipemic Healthy Male Subjects (Parallel Group Comparison, Randomized, Placebo Controlled, Partly Double Blind [Pravastatin Open])
Brief Title: Pharmacodynamics, Preliminary Pharmacokinetics and Tolerability of BIBB 1464 (Tablet) in Hyperlipemic Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1178.2
Record Dates: First submitted 2014-08-28; First posted 2014-09-01 (Estimated); Last update posted 2014-09-01 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Pravastatin

ARMS (5):
- BIBB 1464 MS low dose (Experimental)
  Interventions: Drug: BIBB 1464 MS low dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Pravastatin (Active Comparator)
  Interventions: Drug: Pravastatin
- BIBB 1464 MS medium dose (Experimental)
  Interventions: Drug: BIBB 1464 MS medium dose
- BIBB 1464 MS high dose (Experimental)
  Interventions: Drug: BIBB 1464 MS high dose

INTERVENTIONS:
Drug: BIBB 1464 MS low dose
  Arms: BIBB 1464 MS low dose
Drug: Placebo
  Arms: Placebo
Drug: Pravastatin
  Arms: Pravastatin
Drug: BIBB 1464 MS medium dose
  Arms: BIBB 1464 MS medium dose
Drug: BIBB 1464 MS high dose
  Arms: BIBB 1464 MS high dose

SUMMARY:
Lipid lowering effect, investigation of pharmacodynamics (inhibition of oxidosqualene cyclase, monoepoxysqualene (MES) as marker), safety / tolerability and preliminary pharmacokinetics

ELIGIBILITY:
Inclusion Criteria:

* Healthy male Caucasian subjects as determined by results of screening
* Written informed consent in accordance with GCP and local legislation given
* Age >= 18 and <= 65 years
* Broca >= - 20% and <= + 30%
* LDL-cholesterol level >= 3.3 mmol/L at pre-screening and at the two screening visits

Exclusion Criteria:

* Any finding of the medical examination. (including blood pressure, pulse rate and ECG) deviating from normal and of clinical relevance
* Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal (including thyroid) disorder
* Surgery of the gastro-intestinal tract (except appendectomy)
* Disease of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
* History or orthostatic hypotension, fainting spells or blackouts
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged the investigator
* Intake of drugs with a long half-life (> 24 hours) (<= 1 month prior to administration or during the trial)
* Use of any drugs which might influence the result of the trial (<= 10 days prior to administration or during the trial)
* Participation in another trial with an investigational drug (<= 2 month prior to administration or during the trial)
* Smoker (> 10 cigarettes or > 3 cigars or >3 pipes/day)
* Inability to refrain from smoking during the period of the study
* Alcohol abuse (>60/g/day)
* Drug abuse
* Blood donation (>400ml <=1 month prior to administration)
* Excessive physical activities (<=5 days prior to administration)
* Any laboratory value outside the normal range of clinical relevance
* LDL - cholesterol screening measurements day -1 and day -7 the different between these two values exceed 12% of the higher dose
* subjects who are vegetarian

Eye-lens

* Cataract extraction in one or both eyes deemed likely within 2 years ("senile", non-idiopathic will not automatically exclude patients from participation)
* Lens Opacities Classification System (LOCS) III grade >3.0 (for nuclear opalescence or cortical grad) >0.5 (for posterior sub capsular grad)
* Log MAR Bailey-Lovie visual acuity >0.5
* Corneal or conjunctival problems which would preclude lens photography
* Shallow anterior chamber with risk of angle-closure glaucoma
* Pupil will not dilate to at least 6 mm
* Visually significant fundus pathology in clinician's judgment
* Amblyopia, optic nerve disease, iritis, history of eye surgery, argon or YAG laser, major eye trauma, extended use (daily for >3 month) of ocular or systemic corticosteroid treatment , use of anticoagulants, or glaucoma therapy, or participation in another clinical trial investigation an anti-cataract or cataractogenic formulation within the last year

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2000-01; Primary Completion 2000-05 (Actual)

PRIMARY OUTCOMES:
Percentage change of LDL plasma cholesterol | baseline, 2 weeks
Percentage change of total plasma cholesterol | baseline, 2 weeks

SECONDARY OUTCOMES:
Percentage change in lipid profile | baseline, 1 week
Number of patients with adverse events | Up to day 42
Number of patients with clinical significant findings in eye lens opacification | Up to day 42
Number of patients with clinical significant findings in laboratory parameters | Up to day 28
Number of patients with clinical significant findings in electrocardiogram (ECG) | Up to day 28
Number of patients with clinical significant findings in physical examination | Up to day 28
Number of patients with clinical significant findings in vital signs | Up to day 15
Investigator assessed tolerability on a 4 point scale | day 42
Amount of drug excreted in urine | Up to day 15
Drug plasma concentration | Up to day 28
Monoepoxysqualene (MES) plasma concentration | Up to day 28